CLINICAL TRIAL: NCT06171958
Title: Cohort Study of Intravenous Contrast-media Influence on Decreased Renal Function
Brief Title: Incidence of Acute Kidney Injury After Administration of Iodine Contrast Media in Patients With Reduced Renal Function
Acronym: COINCIDES
Status: Recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: COINCIDES
Record Dates: First submitted 2023-11-16; First posted 2023-12-15 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Acute Kidney Injury Following Administration of Contrast Media
Keywords: cohort study; incidence study; acute kidney injury; contrast media; tomography, x-ray computed
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICM: Patients receiving ICM at CT
  Interventions: Drug: Iodine-containing Contrast Media
- No ICM: Patients not receiving ICM at CT

INTERVENTIONS:
Drug: Iodine-containing Contrast Media — Patients will receive or not receive ICM depending on their medical need.
  Groups: ICM

SUMMARY:
This study is examining if injection of iodine contrast media increases the risk of acute kidney injury in patients with severely reduced renal function. All patients who have a medical need for a computerized tomography, either with or without iodine contrast media, and has a renal function of less than estimated glomerular filtration rate (eGFR) 30 will be recruited. Blood and urine samples will be collected at baseline, three and 21 days after the computerized tomography. Additionally, we will examine if the decision to use iodine contrast media or not was easy or difficult if the use of iodine contrast media potentially changed the patient care and if it might have been lifesaving.

DETAILED DESCRIPTION:
This is a single centre prospective cohort study performed at a tertiary level, university hospital in Sweden.

Background data included age, sex, height, and weight. Body surface area (BSA) is calculated with DuBois formula. Clinical history consists of chronic heart failure (CHF), chronic kidney disease (CKD), diabetes mellitus (DM), hypertension and liver failure. Details regarding the CT such as examined body part, clinical question on CT referral, if iodine contrast media (ICM) was used and, if so, which dose, type and concentration is going to be recorded.

Blood and urine samples will be collected three times prospectively and, if available, previously recorded plasma creatinine values will be recorded once as well. The retrospective value is recorded at least seven days before CT. The prospective values are going to be recorded within 24 hours before CT, 72 hours after CT and 21 days after CT. The following biomarkers are analysed in plasma: bicarbonate, creatinine, cystatin C and endostatin. The following biomarkers are analysed in urine: angiotensinogen (AGT), creatinine, cystatin C, endostatin, kidney injury molecule-1 (KIM-1), neutrophile gelatinase associated lipase (NGAL) and tissue inhibitor of metalloproteinase-2 (TIMP-2). The revised Lund-Malmö formula is used to calculate eGFR based on creatinine. The Caucasian and Asian Paediatric and Adult subjects (CAPA) formula is used to calculate eGFR from Cystatin C.

Five yes or no-questions are going to be answered, two before the exam and three after. The questions answered before the exam will be answered by the radiologist who decided upon the exam protocol, and they are investigating if the decision to use ICM or not was easy to make. The questions after the exam are going to be answered by two senior radiologists independent of each other and they relate to if ICM helped in the discovery of clinically relevant information and if that information/condition was life-threatening. The third question will be answered by going through the patient's discharge summary and is looking at the main diagnosis and if that diagnosis would have been easier to discover with the use of ICM. Since no clear definition of life-threatening exists all diagnoses that were considered life-threatening will be stated in the manuscript. The data will be recorded in the electronic data capture REDCap.

Sample size has been calculated based on an incidence of 14%, a margin of error of 5% and a 95% confidence interval. If there will be to much missing data to run a complete observation analysis, and especially if it is unbalanced between ICM and no ICM an imputation will be performed.

Association will be evaluated with logistic regression. Test of difference among groups will be performed with chi-2 test for categorical variables and the Kruskal-Wallis test for continuous variables. If to many data points are missing and especially if it is unbalanced between groups imputation will be performed. Data will be presented as median and interquartile range or as frequency in percent where suitable. A significance level of 0.05 will be used.

ELIGIBILITY:
Inclusion Criteria:

* eGFR <30 mL/min/1.73m2, calculated with the revised Lund-Malmö formula and plasma creatinine.
* Medical need of either an ICM-enhanced or unenhanced CT

Exclusion Criteria:

* <18 years of age
* Ongoing renal replacement therapy
* Ongoing treatment with nephrotoxic drugs. Drugs classified as nephrotoxic are acyclovir, aminoglycosides, ciclosporins, cisplatin, methotrexate, non-steroidal anti-inflammatory drugs (except low-dose aspirin) and vancomycin administered intravenously.
* Known allergy to ICM who and have not received prophylactic treatment (if patient belongs to ICM arm)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients referred for a CT at Uppsala University Hospital which is a tertiary level hospital that also handles most emergency cases in Uppsala county, Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-contrast acute kidney injury (PC-AKI) | This outcome is measured 72 hours after CT.
  The primary outcome, PC-AKI, is defined and staged according to the creatinine-based criteria from Kidney Disease Improve Global Outcome (KDIGO) [5]. If any of these criteria are fulfilled 72 hours after ICM administration the patient had PC-AKI. The urine output criterion was not used in this study. PC-AKI should be read as post-CT AKI in patients not receiving ICM.
Incidence of long-term decline in renal function | This outcome is measured 21 days after CT.
  Any remaining increase in creatinine compared to baseline.
Incidence of long-term decline in renal function | This outcome is measured 21 days after CT.
  Any remaining increase in cystatin C compared to baseline.

SECONDARY OUTCOMES:
Incidence of mortality | 21 days
  Mortality will be recorded during the follow-up period.
Incidence of need for renal replacement therapy | 21 days
  A need for any form of renal replacement during the follow-up period.

OTHER OUTCOMES:
Incidence of elevated plasma bicarbonate | Data will be recorded at 72 hours and 21 days.
  Elevation of bicarbonate in plasma compared with baseline value.
Incidence of elevated plasma endostatin compared to baseline | Data will be recorded at 72 hours and 21 days.
  Elevation of endostatin in plasma compared with baseline value.
Incidence of elevated urine endostatin | Data will be recorded at 72 hours and 21 days.
  Elevation of endostatin in urine compared with baseline value.
Incidence of elevated urine creatinine | Data will be recorded at 72 hours and 21 days.
  Elevation of creatinine in urine compared with baseline value.
Incidence of elevated urine cystatine C | Data will be recorded at 72 hours and 21 days.
  Elevation of cystatine C in urine compared with baseline value.
Incidence of elevated urine KIM-1 | Data will be recorded at 72 hours and 21 days.
  Elevation of KIM-1 in urine compared with baseline value.
Incidence of elevated urine NGAL | Data will be recorded at 72 hours and 21 days.
  Elevation of NGAL in urine compared with baseline value.
Incidence of elevated urine TIMP-2 | Data will be recorded at 72 hours and 21 days.
  Elevation of TIMP-2 in urine compared with baseline value.

CONTACTS AND LOCATIONS:
Locations (1):
- Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analysed during the current study are not publicly available due national and European Union regulations regarding patient related data but are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Du BOIS D, Du BOIS EF. CLINICAL CALORIMETRY: TENTH PAPER A FORMULA TO ESTIMATE THE APPROXIMATE SURFACE AREA IF HEIGHT AND WEIGHT BE KNOWN. Archives of Internal Medicine. 1916;XVII(6_2):863-71.
- [Background] Bjork J, Grubb A, Sterner G, Nyman U. Revised equations for estimating glomerular filtration rate based on the Lund-Malmo Study cohort. Scand J Clin Lab Invest. 2011 May;71(3):232-9. doi: 10.3109/00365513.2011.557086. Epub 2011 Mar 10. PMID 21391777
- [Background] Grubb A, Horio M, Hansson LO, Bjork J, Nyman U, Flodin M, Larsson A, Bokenkamp A, Yasuda Y, Blufpand H, Lindstrom V, Zegers I, Althaus H, Blirup-Jensen S, Itoh Y, Sjostrom P, Nordin G, Christensson A, Klima H, Sunde K, Hjort-Christensen P, Armbruster D, Ferrero C. Generation of a new cystatin C-based estimating equation for glomerular filtration rate by use of 7 assays standardized to the international calibrator. Clin Chem. 2014 Jul;60(7):974-86. doi: 10.1373/clinchem.2013.220707. Epub 2014 May 14. PMID 24829272
- [Background] McDonald JS, McDonald RJ, Carter RE, Katzberg RW, Kallmes DF, Williamson EE. Risk of intravenous contrast material-mediated acute kidney injury: a propensity score-matched study stratified by baseline-estimated glomerular filtration rate. Radiology. 2014 Apr;271(1):65-73. doi: 10.1148/radiol.13130775. Epub 2014 Jan 16. PMID 24475854
- [Background] KDIGO. KDIGO Clinical Practice Guideline for Acute Kidney Injury. Kidney International, Supplements. 2012;2(1).